CLINICAL TRIAL: NCT02380859
Title: Treatment of Gait Disturbance in Parkinson's Disease With Prism Adaptation
Brief Title: Prism Adaptation Treatment of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Stephen L. Lee, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D15047
Record Dates: First submitted 2015-02-24; First posted 2015-03-05 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Parkinson
Keywords: problems of gait and balance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prism adaptation (Active Comparator): Patients will undergo twice daily adaptation to upward shifts in vision. Participants will be provided with goggles fitted with prismatic lenses that shift vision upward by 25 dioptres (about 17 degrees). While wearing the lenses, participants point to two 10cm-diameter visual targets positioned one above the other (about 20cm apart) on a wall, returning their pointing arm to their chest between each pointing movement. Participants make 50 pointing movements, as fast and as accurately as possible. Such a procedure induces a downward sensorimotor adaptation of pointing movements. Participants undergo this training twice a day (morning and evening) for two weeks in a self-guided fashion.
  Interventions: Behavioral: Prism adaptation
- Sham adaptation (Sham Comparator): Participants undergo the same treatment protocol as described in the active comparator arm, with the exception that they wear goggles fitted with neutral lenses that do not induce sensorimotor adaptation.
  Interventions: Behavioral: Prism adaptation

INTERVENTIONS:
Behavioral: Prism adaptation — Prism adaptation is one type of sensorimotor adaptation. Prism adaptation described any adaptation to a prismatic shift in vision (i.e. any magnitude or direction of shift). In this study we are using adaptation to upward-shifting prisms, which induces a downward sensorimotor after-effect.
  Other Names: sensorimotor adaptation, visual adaptation

SUMMARY:
Subjects diagnosed with Idiopathic Parkinson's Disease, between ages of 40-85 inclusive, who have been referred for gait training. Since there can be subtle differences in the brain organization of left- and right-handed people that may influence some of the measurements, right handed participants are preferred. However, a left handed participant may be considered. Participants will be randomly assigned to one of two groups to undergo two weeks of twice-daily sessions. Group A receiving goggles fitted with lenses that distort vision and Group B patients receiving sham goggles

DETAILED DESCRIPTION:
The participants will be trained to undergo two daily sessions of visual adaptation at home for 14 consecutive days. For each adaptation session, subject will sit in a chair within reaching distance of a wall or cabinet upon which two dime-sized targets will be placed (one above the other, approximately ten inches apart). While wearing goggles, you will point rapidly to one target then the next, bringing the hand back to his/her torso between each pointing movement. They will be instructed to perform these movements "as quickly as possible" for a total of 50 pointing movements in each treatment session. After performing the 50 pointing movements, they will remove their goggles. Throughout the treatment period they will be asked to keep a diary in which they will log the time and duration of each prism adaptation session. At the first and second site visits, participants will be assessed for posture, gait and activities of daily living which will include some questionnaires. Questionnaires will be sent via mail after post-treatment at one week,1 month and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease
* Referral for gait training
* Aged 40 -85
* If the subject is taking CNS-acting medications (benzodiazepines, hypnotics, antidepressants), regimen must be stable for 30 days prior to baseline visit
* Subjects with Stage 11.5 - Stage IV (Hoehn and Yahr scale) where stage II.5 is bilateral involvement with axial involvements, but without balance difficulty, to Stage IV where one has severe disability but is still able to walk or stand unassisted
* Subjects with any of the following abnormal scores (greater than 0) in the MDS-UPDRS Part III; a) Part III.10 Gait; b) Part III.11 Freezing of gait c) Part III.12 Postural Stability; subjects with Timed up and go test >12 seconds
* Right handed participants are preferred due to the cortical lateralization of functions related to sensorimotor adaptation and postural control.
* However, we will recruit left-handed participants if there are insufficient right-handed volunteers.

Exclusion Criteria:

* Subjects with a known psychiatric comorbidity that in the investigator's opinion would compromise participation in the study; subjects with a neurologic diagnosis, other than Parkinson's disease that can cause imbalance and gait impairment (e.g., multiple sclerosis, stroke, subdural hematoma, peripheral neuropathy)
* Injury or impairment to the right arm (other than that which is due to Parkinson's disease) that would affect pointing movements; subjects with normal score on UPDRS part III
* Classified as legally blind or lacking sufficient visual acuity to view the target and pointing hand during prism adaptation
* Lacking sufficient understanding of verbal and written information in English to complete any of the consent screening forms.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2017-07 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L. Lee, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Darmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bultitude JH, Pidgeon DM, LeBlanc PR, Jeffreys CA, Alexandre FP, Lee SL. Two weeks of twice-daily prism adaptation treatment does not improve posture or gait in Parkinson's disease: a double-blind randomized controlled trial. Trials. 2021 Nov 25;22(1):846. doi: 10.1186/s13063-021-05832-2. PMID 34823572

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a protocol violation in our intended randomization procedure in that participants were randomized to treatment or control groups with replacement instead of without replacement. This resulted in uneven group numbers, rather than the equal group numbers that was intended.
Groups:
- Real Prism Adaptation: Participants were randomized to undergo treatment that involved adaptation to 15º upward shifts in vision.
- Sham Prism Adaptation: Participants were randomized to placebo lenses that distorted vision without vertical shift.
Period: Overall Study
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Started | 19 | 13
Completed | 17 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Real Prism Adaptation: Participants were randomized to treatment prisms, designed to shift vertical orientation slightly by 1.5 degrees
- Total: Total of all reporting groups
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.7) | 68.3 (8.2) | 69.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 12 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 13 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Postural Control - Reaction Time on the Limits of Stability Test (Smart Equitest Balance Master System)
Description: The participant stood on the platform in front of a monitor. Nine squares were presented on the monitor representing locations relative to the upright starting position: one in the centre of the screen (upright) and the remaining eight forming an ellipse around the central square. The participant's COG was indicated on the screen by the position of a stick figure avatar. At the beginning of each trial the participant was instructed to stand upright, keeping the COG cursor over the central target. A circular target appeared in one of eight other targets. The participant was required to move the COG cursor towards the second target as quickly and as accurately as possible by leaning their body while keeping their feet in the same location, and to then hold a position as close to the target as possible. Reacting times were recorded for 8 trials per location. Mean change (post-pre) in seconds
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
Seconds | 0.09 (0.29) | -0.02 (0.36)

2. Primary Outcome: Change in Postural Control - Maximum Velocity on the Limits of Stability Test (Smart Equitest Balance Master System)
Description: The participant stood on the platform in front of a monitor. Nine squares were presented on the monitor representing locations relative to the upright starting position: one in the centre of the screen (upright) and the remaining eight forming an ellipse around the central square. The participant's COG was indicated on the screen by the position of a stick figure avatar. At the beginning of each trial the participant was instructed to stand upright, keeping the COG cursor over the central target. A circular target appeared in one of eight other targets. The participant was required to move the COG cursor towards the second target as quickly and as accurately as possible by leaning their body while keeping their feet in the same location, and to then hold a position as close to the target as possible. Maximum velocity was recorded for 8 trials per location.
Time Frame: Baseline (Day 0) and Day 15
Population: Average change time; mean change (post-pre) meters per second
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
meters per second | 0.54 (0.67) | 0.11 (0.62)
Statistical Analysis 1: Comparison: Real Prism Adaptation vs Sham Prism Adaptation; Group (real, sham) x Time (pre, 1d post) x Stepping Direction (forward, backward) ANOVA; Test type: Superiority; p = 0.005, ANOVA

3. Primary Outcome: Change in Postural Control - Maximum Extension on the Limits of Stability Test (Smart Equitest Balance Master System)
Description: The participant stood on the platform in front of a monitor. Nine squares were presented on the monitor representing locations relative to the upright starting position: one in the centre of the screen (upright) and the remaining eight forming an ellipse around the central square. The participant's COG was indicated on the screen by the position of a stick figure avatar. At the beginning of each trial the participant was instructed to stand upright, keeping the COG cursor over the central target. A circular target appeared in one of eight other targets. The participant was required to move the COG cursor towards the second target as quickly and as accurately as possible by leaning their body while keeping their feet in the same location, and to then hold a position as close to the target as possible. Maximum extension of the COG over the feet was recorded for 8 trials per location.
Time Frame: Baseline (Day 0) and Day 15
Population: Average change in Maximum Extension between baseline and day 15
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
meters | 3.0 (9.8) | 0.63 (10.4)

4. Primary Outcome: Change in Postural Control - Composite Score on the Sensory Organisation Test SMART EquiTest Balance Master
Description: The participant is asked to maintain an upright posture under six different conditions of sensory feedback:
  * Condition 1:Normal vision, fixed support
  * Condition 2:Absent vision, fixed support
  * Condition 3:Sway-referenced vision, fixed support
  * Condition 4:Normal vision, sway-referenced support
  * Condition 5:Absent vision, sway-referenced support
  * Condition 6:Sway-referenced vision, sway-referenced support
  The equilibrium score for each condition compares the subject's anterior/posterior (AP) sway during each trial to the theoretical sway stability limit of 12.5 degrees. A composite equilibrium score (0-100, higher score indicates better outcome) quantifies the overall COG sway or postural stability across the sensory conditions and is calculated by:
  * Independently averaging the score for conditions 1 and 2;
  * Adding these two scores to the equilibrium scores from each trial of sensory conditions 3, 4, 5, and 6; and
  * Dividing that sum by the total number of trials.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: change in percentage
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
change in percentage | 4.3 (9.2) | 2.5 (10.4)

5. Secondary Outcome: Change in Gait - Step Length on the Walk Across Test (SMART Equitest Balance Master)
Description: The WA quantifies characteristics of gait as the patient walks across the length of the force plate. The test characterizes steady state gait by having the patient begin well behind and continuing beyond the force plate. Measured parameters are average step width, average step length, speed and step length symmetry.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
cm | -3.0 (30.4) | -4.1 (32.6)

6. Secondary Outcome: Change in Gait - Step Speed in the Walk Across (SMART Equitest Balance Master)
Description: as for outcome 5
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
cm/s | 5.0 (19.5) | 1.3 (22.0)

7. Secondary Outcome: Change in Gait - Timed Up and Go Task
Description: Timed Up and Go Test (TUG). Patients are seated in a chair and instructed to stand up, walk three meters, turn around, walk back, and sit down. The time (in seconds) is recorded.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
seconds | -1.8 (4.8) | -0.25 (1.3)

8. Secondary Outcome: Change in Gait - Functional Gait Assessment
Description: Functional Gait Assessment. This 10-item test assesses dynamic balance and postural stability during gait. Items consist of specific walking tasks such as stepping over an obstacle, changing speed of walking upon the assessor's instruction, and walking backwards. The assessor scores the patient's performance from 0 ("severe impairment") to 3 ("normal") and a total is calculated out of 30.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
scores on a scale | 1.8 (4.8) | 1.0 (1.7)

9. Other Pre Specified Outcome: Change in Activities of Daily Living - New Freezing of Gait
Description: Average change in score relating to new freezing of gate utilizing the New Freezing of Gait Questionnaire. This nine-item questionnaire detects and evaluates the impact and severity of freezing of gait on locomotion and daily activities. Items are scored from 0 or 1 to 3 or 4, with higher numbers indicating greater impact and severity. A total score out of 28 is calculated.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
scores on a scale | -0.19 (4.19) | -5.0 (1.40)

10. Other Pre Specified Outcome: Change in Activities of Daily Living - Falls Efficiency
Description: Average change in score evaluated using the Falls Efficiency Scale. This ten-item questionnaire asks people to rate their confidence in performing daily activities without falling. Responses are given on a scale from 0 ("very confident") to 10 ("not very confident") and a total score out of 100 is computed.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
scores on a scale | 2.16 (10.11) | -10.70 (2.97)

11. Other Pre Specified Outcome: Change in Activities of Daily Living - Activity-specific Balance Confidence Scale
Description: Activities-specific Balance Confidence Scale. This 16-item questionnaire is similar to the Falls Efficiency Scale, but has greater sensitivity to gait impairments in more ambulatory patients. Responses are given on a scale from 0 ("very confident") to 10 "not very confident") and a total score out of 100 is computed.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
scores on a scale | -0.57 (10.7) | -5.8 (12.8)

12. Other Pre Specified Outcome: Change in Activities of Daily Living - Parkinson's Disease Questionnaire
Description: Parkinson's Disease Questionnaire (PDQ-39), mobility and activities of daily living sections. This 39-item questionnaire is the most widely-used Parkinson's Disease specific measure of health and daily function. Participants indicate the extent to which they have experienced problems with different aspects of mobility and self-care. Each item is scored from 0 ("never have problems") to 4 ("always have problems"), and a percentage is calculated. In addition to the total score, the mobility (questions 1-10) and activities of daily living (questions 11-16) sub-sections can be analysed separately to assess changes in these specific outcomes. The responses are summed and scored as a percentage. We analysed the percentage scores for the mobility sub-section, the activities of daily living sub-section, and the total percentage. Higher values indicate worse outcome.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
percentage
  Mobility subscale (%) | -0.89 (8.83) | -2.50 (13.27)
  Activities of daily living subscale (%) | -0.63 (12.48) | 3.8 (11.2)
  Total (%) | 0.21 (6.13) | 1.78 (8.27)

13. Primary Outcome: Change in Postural Control - Forward-backward Displacement of Centre of Gravity on the Sensory Organisation Test SMART EquiTest Balance Master
Description: The participant is asked to maintain an upright posture under different conditions of sensory feedback. Proprioceptive feedback to the feet and joints is manipulated by allowing the platform to tilt to directly follow the participant's anteroposterior body sway (constant proprioception) or by maintaining the standing platform in a fixed horizontal position (normal proprioceptive feedback). Visual feedback is provided by asking the participant to close their eyes (no visual feedback), asking the participant to open their eyes and allowing the visual surround to tilt directly following the participant's anterioposterior body sway (constant visual feedback), or by asking the participant to keep their eyes open and maintaining the visual surround in a fixed position (normal visual feedback). Forward-backward displacement of COG is recorded in degrees.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
Degrees | 0.05 (1.3) | -0.12 (0.62)

14. Primary Outcome: Change in Postural Control - Composite Latency Score on the Motor Control Test
Description: The MCT assesses the ability of the automatic motor system to quickly recover following an unexpected external disturbance. Sequences of small, medium or large platform translations (scaled to the patient's height) in forward and backward directions elicit automatic postural responses. Translation of the surface in one horizontal direction results in displacement of the COG away from center in the opposite direction relative to the base of support. To restore normal balance, a quick movement of the COG back to the center position is required. A composite latency value is provided as the time in milliseconds between the force plate translation and the patient's active corrective responses, averaged across all translation sizes and directions.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
ms | 1.9 (13.6) | 2.1 (23.1)

15. Primary Outcome: Change in Postural Control - Composite Latency Score on the Berg Balance Scale
Description: Berg Balance Scale. This 14-item test assesses balance during different tasks. Items consist of specific items such as standing with eyes closed, retrieving an object from the floor, and turning to look behind. The assessor rates the patient's performance from 0 ("lowest level of function") to 4 ("highest level of function") and a total is calculated out of a maximum score of 56.
Time Frame: Baseline (Day 0) and Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
Number analyzed (Participants) | 17 | 13
scores on a scale | 0.38 (2.4) | -0.69 (2.4)

ADVERSE EVENTS:
Time Frame: From consent until study completion, approximately 3 months.
Arm/Group | Real Prism Adaptation | Sham Prism Adaptation
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 1/17 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Prism Adaptation (N=17) | Sham Prism Adaptation (N=13)
Concusion (Nervous system disorders) | 0 (0) | 1 (1)
Freezing (Nervous system disorders) | 1 (1) | 0 (0) — Foot Froze and balance was affected
Blurry Vision/Dizzy (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT02380859/Prot_SAP_000.pdf